CLINICAL TRIAL: NCT00314860
Title: A 12-Week, Randomized, Double-Blind, Parallel Group, Multicentre Study to Assess the Tolerability and Clinical Benefits of Ropinirole Extended Release (XR) Tablets Compared With Ropinirole Immediate Release (IR) Tablets in Subjects With Restless Legs Syndrome (RLS)
Brief Title: RLS In Adults: Comparing Immediate Release Formulation With Extended Release Formulation Of Ropinirole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101468/204
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Restless Legs Syndrome; Restless Legs Syndrome (RLS)
Keywords: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ropinirole Extended Release (XR)

SUMMARY:
Restless Legs Syndrome (RLS) study in adults comparing immediate release ropinirole with extended release ropinirole over 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary RLS according to RLS Diagnostic Clinical Interview and International Restless Legs Syndrome Study Group Diagnostic Criteria.
* Disturbed sleep, with both evening (between 5:00 pm and 8:00 pm) and night time (between 8:00 pm and 8:00 am) symptoms requiring treatment.

Exclusion criteria:

* Signs of secondary RLS.
* Primary sleep disorder or movement disorder other than RLS.
* Unstable medical conditions.
* Inability to tolerate dopamine agonists or dopamine antagonists.
* Unwilling to discontinue any medications currently being taken to treat RLS symptoms.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2006-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate the superior tolerability of ropinirole extended release compared to ropinirole immediate release in adult subjects with RLS requiring evening and night-time coverage of RLS symptoms | 12 Weeks

SECONDARY OUTCOMES:
To compare the safety profile and to evaluate the clinical benefits (as assessed by efficacy endpoints and patient-reported outcomes) of ropinirole extended release compared to ropinirole immediate release in subjects with RLS. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (88):
- United States (28):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Burlingame, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Winnetka, California
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, West Yarmouth, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Burlington, Vermont
- Australia (3):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
- Austria (2):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Liège
- Denmark (4):
  - GSK Investigational Site, Glostrup Municipality
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Koebenhavn NV
  - GSK Investigational Site, Odense C
- France (9):
  - GSK Investigational Site, Anzin
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Montbrison
  - GSK Investigational Site, Nancy
  - GSK Investigational Site, Pessac
- Germany (6):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Köthen, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Gera, Thuringia
- Italy (5):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Pisa, Tuscany
- Netherlands (7):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Geldermalsen
  - GSK Investigational Site, Grubbenvorst
  - GSK Investigational Site, Hoogwoud
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Roelofarendsveen
  - GSK Investigational Site, Zwolle
- Norway (3):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Sandvika
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Zaragoza
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Helsingborg
  - GSK Investigational Site, Örebro
- United Kingdom (8):
  - GSK Investigational Site, Chesterfield, Derbyshire
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Frome, Somerset
  - GSK Investigational Site, Coventry, Warwickshire
  - GSK Investigational Site, Trowbridge, Wiltshire
  - GSK Investigational Site, Corsham
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Ledbury

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 101468/204 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 101468/204 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 101468/204 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 101468/204 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 101468/204 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101468/204 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 101468/204 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register